CLINICAL TRIAL: NCT06831773
Title: Phase II Clinical Study of Carbon Ion Combined with Photon Radiotherapy for High-grade Glioma
Brief Title: Clinical Study of Carbon Ion Radiotherapy for High-grade Glioma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gansu Wuwei Tumor Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 185647
Record Dates: First submitted 2025-02-05; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Carbon Ion Radiotheray; High-grade Glioma; Heavy Ion Radiotherapy
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Intervention Model Description: Carbon ion combined with photon radiotherapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study group (Experimental): PTV1 was firstly treated with photon radiotherapy (started within 30 days after surgery), with a total dose of 50Gy for 25 times. After photon radiotherapy, PTV2 carbon ion radiotherapy was started, the total dose was 24.8Gy(RBE), 8 times. 3.1Gy(RBE)/fx; 1fx/ day, 5 days/week
  Interventions: Radiation: Carbon ion combined with photon radiotherapy

INTERVENTIONS:
Radiation: Carbon ion combined with photon radiotherapy — PTV1 was first treated with photon radiotherapy (started within 30 days after surgery), with a total dose of 50Gy, 25 times; After photon radiotherapy, PTV2 carbon ion radiotherapy was started, the total dose was 24.8Gy(RBE), 8 times. 3.1Gy(RBE)/fx; 1fx/ day, 5 days/week.

SUMMARY:
The objective is to use the advantages of heavy ion physical dosimetry and biology to improve the tumor control rate and long-term survival rate of high-grade glioma, reduce the occurrence of brain tissue radiation damage caused by increasing prescription dose, and provide new treatment suggestions for glioma radiotherapy.

DETAILED DESCRIPTION:
The investigators tend to make reference to the prescribed dose and segmentation method in the phase I/II clinical study program completed by Mizoe et al., NIRS. It is estimated that the 1-year OS rate of high-grade glioma treated with photon (50Gy divided into 25 times) followed by carbon ion push (24.8GyE divided into 8 times) can reach 87.8%, and the target value is set at 61.1%. A single-center, single-arm, prospective Phase II clinical trial was conducted to evaluate the safety and efficacy of this regimen. The primary end points were treatment-related toxicity, dose-restricted toxicity, and progression-free survival, while the secondary end points were survival and objective response rate. A safe and effective segmentation dose for high-grade glioma suitable for the investigators' facility and RBE model was obtained. Using the physical dosimetry and biological advantages of heavy ions, the investigators can improve the tumor control rate and reduce the occurrence of radiation damage in peripheral brain tissue caused by increasing prescription dose, and provide new treatment suggestions for glioma radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥14 years and ≤80 years;
2. Indications: According to the criteria of the 5th edition of WHO Classification of Central Nervous System Tumors published in 2021, histological characteristics and molecular phenotype were integrated, and the molecular phenotype was IDH wild-type glioma and IDH mutant WHO Grade Ⅲ and Ⅳ glioma. They mainly include: IDH wild-type low-grade glioma (Grade 4 astrocytoma according to the 2021 WHO classification definition); Anaplastic Astrocytoma, AA; anaplastic astrocytoma, AA; Anaplastic Oligodendroglioma, AOG; anaplastic oligodendroglioma, AOG; Anaplastic Oligoastrocytoma, AOA; anaplastic oligoastrocytoma, AOA; Glioblastoma Multiforme, GBM. Regardless of surgical completeness, i.e. after total, subtotal, or partial resection, and after stereotactic or craniotomy.
3. No distant or intraspinal spread and metastasis; A single or two intracranial lesions may be covered by the same radiotherapy plan.
4. The treatment conditions before this radiotherapy were as follows: First radiotherapy: no interventional, photodynamic or other tumor ablation was performed within 4 weeks before this radiotherapy; The operative wound has fully healed.
5. Can accept MRI and enhanced CT examination, and there are no metal artifacts in CTV;
6. No history of other malignant tumors (except cured skin cancer and stage 0 cervical cancer);
7. Liver function, kidney function and bone marrow function were basically normal (ALT and AST < 1.5 times of high normal value (ULN), bilirubin < 1.5×ULN; Adult endogenous creatinine clearance rate of 60ml/min or serum creatinine SCR≤140μmoI/L, BUN≤6.8mmol/L; Hemoglobin level >9 g/dL; White blood cell count ≥3.0*109/L; Platelet count ≥100*109/L;)
8. Good physical condition, i.e. ECOG (Eastern United States Oncology Collaboration Group) 0~2; There were no complications such as severe pulmonary hypertension, cardiovascular disease, peripheral vascular disease, and severe chronic heart disease that may affect radiotherapy. Cardiac function grade 1. (According to the New York College of Cardiology Cardiac Function Scale (NYHA)
9. Adequate functions of major organs;
10. Predicted survival (after treatment) ≥6 months;
11. Informed consent has been signed by the patient or his legal representative before radiotherapy.

Exclusion Criteria:

1. WHOII-IV glioma unconfirmed by pathology;
2. Patients who cannot lie still for 30 minutes;
3. Secondary treatment of recurrent tumors
4. There have been distant metastases, or scattered or multiple (>2) intracranial lesions;
5. Have received conventional photon/proton/carbon ion radiotherapy to the head;
6. Have received intracranial radioactive particle implantation with metal implants that may affect the dose of particle radiation therapy;
7. Unable to receive MRI with claustrophobia or a pacemaker or metal implant
8. Pacemakers or other metal implants that may be interfered with normal function by high-energy radiation or may affect the dose of radiation target;
9. The dose limit for organs at risk cannot reach the preset safe dose limit
10. Pregnancy (confirmed by serum or urine β-HCG test) or lactation
11. losing more than 20% of your body weight within six months;
12. Persons with AIDS, including those who have received antiretroviral therapy; Active stage of syphilis;
13. Accompanied by serious comorbiditions, including uncontrolled systemic or co-existing diseases (pulmonary insufficiency, cardiovascular, pulmonary, liver, kidney, diabetes, etc.), drug or alcohol abuse, dependence, addiction, and/or mental illness that prevent the successful implementation of the trial protocol;
14. Patients with poor compliance, including those who may not be able to complete the treatment plan or receive prescribed follow-up and examination;
15. have had other malignant neoplasms (except cured skin cancer and stage 0 cervical cancer);
16. There are contraindications to radiotherapy;
17. Participated in other drug clinical trials within 30 days prior to enrollment in this study;
18. having no or limited capacity for civil conduct;
19. Any medical history that, in the investigator's judgment, might interfere with the trial results or increase the patient's risk;
20. Any condition in which the physician considers that participation in the trial is not appropriate, the physician determines that the patient will not benefit from carbon ion radiotherapy, or that there are other co-existing conditions or other factors that may affect carbon ion therapy.
21. Inability to understand the purpose of treatment or unwillingness/inability to sign treatment consent.

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 2 years
  Progression-free survival

SECONDARY OUTCOMES:
overall survival | 2 years
  overall survival
objective remission rate | 2 years
  objective remission rate
Disease control rate | 2 years
  Disease control rate

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojun Li, Study Director — Gansu Wuwei Tumor Hospital
Locations (1):
- Heavy Ion Radiotherapy Department, Wuwei, Gansu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Isono M, Yoshida Y, Takahashi A, Oike T, Shibata A, Kubota Y, Kanai T, Ohno T, Nakano T. Carbon-ion beams effectively induce growth inhibition and apoptosis in human neural stem cells compared with glioblastoma A172 cells. J Radiat Res. 2015 Sep;56(5):856-61. doi: 10.1093/jrr/rrv033. Epub 2015 Jun 11. PMID 26070322
- [Background] Adeberg S, Bernhardt D, Harrabi SB, Uhl M, Paul A, Bougatf N, Verma V, Unterberg A, Wick W, Haberer T, Combs SE, Herfarth K, Debus J, Rieken S. Sequential proton boost after standard chemoradiation for high-grade glioma. Radiother Oncol. 2017 Nov;125(2):266-272. doi: 10.1016/j.radonc.2017.09.040. Epub 2017 Oct 16. PMID 29050959
- [Background] Mizoe JE, Tsujii H, Hasegawa A, Yanagi T, Takagi R, Kamada T, Tsuji H, Takakura K; Organizing Committee of the Central Nervous System Tumor Working Group. Phase I/II clinical trial of carbon ion radiotherapy for malignant gliomas: combined X-ray radiotherapy, chemotherapy, and carbon ion radiotherapy. Int J Radiat Oncol Biol Phys. 2007 Oct 1;69(2):390-6. doi: 10.1016/j.ijrobp.2007.03.003. Epub 2007 Apr 24. PMID 17459607
- [Background] Kong L, Wu J, Gao J, Qiu X, Yang J, Hu J, Hu W, Mao Y, Lu JJ. Particle radiation therapy in the management of malignant glioma: Early experience at the Shanghai Proton and Heavy Ion Center. Cancer. 2020 Jun 15;126(12):2802-2810. doi: 10.1002/cncr.32828. Epub 2020 Mar 13. PMID 32167589
- [Background] Hasegawa A, Mizoe JE, Tsujii H, Kamada T, Jingu K, Iwadate Y, Nakazato Y, Matsutani M, Takakura K; Organizing Committee of the Central Nervous System Tumor Working Group. Experience with carbon ion radiotherapy for WHO Grade 2 diffuse astrocytomas. Int J Radiat Oncol Biol Phys. 2012 May 1;83(1):100-6. doi: 10.1016/j.ijrobp.2011.06.1952. Epub 2011 Nov 19. PMID 22104357
- [Background] Pisapia DJ. The Updated World Health Organization Glioma Classification: Cellular and Molecular Origins of Adult Infiltrating Gliomas. Arch Pathol Lab Med. 2017 Dec;141(12):1633-1645. doi: 10.5858/arpa.2016-0493-RA. PMID 29189064
- [Background] Walker MD, Alexander E Jr, Hunt WE, MacCarty CS, Mahaley MS Jr, Mealey J Jr, Norrell HA, Owens G, Ransohoff J, Wilson CB, Gehan EA, Strike TA. Evaluation of BCNU and/or radiotherapy in the treatment of anaplastic gliomas. A cooperative clinical trial. J Neurosurg. 1978 Sep;49(3):333-43. doi: 10.3171/jns.1978.49.3.0333. PMID 355604
- [Background] Stupp R, Mason WP, van den Bent MJ, Weller M, Fisher B, Taphoorn MJ, Belanger K, Brandes AA, Marosi C, Bogdahn U, Curschmann J, Janzer RC, Ludwin SK, Gorlia T, Allgeier A, Lacombe D, Cairncross JG, Eisenhauer E, Mirimanoff RO; European Organisation for Research and Treatment of Cancer Brain Tumor and Radiotherapy Groups; National Cancer Institute of Canada Clinical Trials Group. Radiotherapy plus concomitant and adjuvant temozolomide for glioblastoma. N Engl J Med. 2005 Mar 10;352(10):987-96. doi: 10.1056/NEJMoa043330. PMID 15758009
- [Background] Stupp R, Hegi ME, Mason WP, van den Bent MJ, Taphoorn MJ, Janzer RC, Ludwin SK, Allgeier A, Fisher B, Belanger K, Hau P, Brandes AA, Gijtenbeek J, Marosi C, Vecht CJ, Mokhtari K, Wesseling P, Villa S, Eisenhauer E, Gorlia T, Weller M, Lacombe D, Cairncross JG, Mirimanoff RO; European Organisation for Research and Treatment of Cancer Brain Tumour and Radiation Oncology Groups; National Cancer Institute of Canada Clinical Trials Group. Effects of radiotherapy with concomitant and adjuvant temozolomide versus radiotherapy alone on survival in glioblastoma in a randomised phase III study: 5-year analysis of the EORTC-NCIC trial. Lancet Oncol. 2009 May;10(5):459-66. doi: 10.1016/S1470-2045(09)70025-7. Epub 2009 Mar 9. PMID 19269895
- [Background] Hegi ME, Diserens AC, Gorlia T, Hamou MF, de Tribolet N, Weller M, Kros JM, Hainfellner JA, Mason W, Mariani L, Bromberg JE, Hau P, Mirimanoff RO, Cairncross JG, Janzer RC, Stupp R. MGMT gene silencing and benefit from temozolomide in glioblastoma. N Engl J Med. 2005 Mar 10;352(10):997-1003. doi: 10.1056/NEJMoa043331. PMID 15758010
- [Background] Gilbert MR, Wang M, Aldape KD, Stupp R, Hegi ME, Jaeckle KA, Armstrong TS, Wefel JS, Won M, Blumenthal DT, Mahajan A, Schultz CJ, Erridge S, Baumert B, Hopkins KI, Tzuk-Shina T, Brown PD, Chakravarti A, Curran WJ Jr, Mehta MP. Dose-dense temozolomide for newly diagnosed glioblastoma: a randomized phase III clinical trial. J Clin Oncol. 2013 Nov 10;31(32):4085-91. doi: 10.1200/JCO.2013.49.6968. Epub 2013 Oct 7. PMID 24101040